CLINICAL TRIAL: NCT04954495
Title: Sexually Transmitted Infections With Mycoplasma Genitalium: Epidemiological, Clinical, Microbiological, Therapeutic Aspects
Acronym: IST_MG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: IST_MG
Record Dates: First submitted 2021-06-21; First posted 2021-07-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Anorectal Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infectious anorectitis is a poorly described clinical entity. Their epidemiology is poorly known, as are their clinical, diagnostic (diagnoses are regularly made in gastroenterology and new diagnostic tools are now available) and therapeutic aspects.

The proctology center of the Marie Thérèse Center is the leading proctology center in the Ile-de-France region both in terms of recruitment and reputation, and drains a large proportion of patients with anorectitis for specialized care. The clinical microbiology laboratory of the Saint Joseph Hospital Group is linked to the Marie Thérèse Center to provide its expertise in the microbiological and infectious aspects of the management of these infections.

In recent years, the analysis of data from this large population of patients referred to the Léopold Bellan proctology center for suspected ano-rectitis has revealed the pathogens Neisseria gonorrhoeae and/or Chlamydia trachomatis.

Mycoplasma genitalium (MG) is an emerging pathogen responsible for Sexually Transmitted Infections (STI) and has been described increasingly in recent years. Studies on this pathogen will allow to better identify risk factors and to target optimized prevention and therapeutic management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patients treated at the Centre de proctologie of the Centre de santé Marie-Thérèse or the GHPSJ (consultation and/or hospitalization) and for whom an anorectal swab will be taken for suspected infectious sexually transmitted ano-rectitis
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patient whose age is ≥ 18 year, treated at the Centre de proctologie of the Centre de santé Marie-Thérèse or the GHPSJ (consultation and/or hospitalization) and for whom an anorectal swab will be taken for suspected infectious sexually transmitted ano-rectitis from June 2021.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-06-17 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical forms of these anorectal infection | Day 1
  This outcome corresponds to the clinical presentation : prevalence of clinical signs [fever (Yes/no), ulcerations (yes/no), purulent proctisis (yes/no), erythematosus proctisis (yes/no), condyloma (yes/no)].

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lourtet, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Price MJ, Ades AE, De Angelis D, Welton NJ, Macleod J, Soldan K, Simms I, Turner K, Horner PJ. Risk of pelvic inflammatory disease following Chlamydia trachomatis infection: analysis of prospective studies with a multistate model. Am J Epidemiol. 2013 Aug 1;178(3):484-92. doi: 10.1093/aje/kws583. Epub 2013 Jun 27. PMID 23813703
- [Background] Vieira VA, Avelino-Silva VI, Cerqueira NB, Costa DA, Costa PR, Vasconcelos RP, Madruga VR, Moreira RI, Hoagland B, Veloso VG, Grinsztejn B, Kallas EG; PrEP Brasil Study Team. Asymptomatic anorectal Chlamydia trachomatis and Neisseria gonorrhoeae infections are associated with systemic CD8+ T-cell activation. AIDS. 2017 Sep 24;31(15):2069-2076. doi: 10.1097/QAD.0000000000001580. PMID 28692536
- See also: Related Info — https://www.ecdc.europa.eu/en/publications-data/chlamydia-control-europe-literature-review